CLINICAL TRIAL: NCT03570827
Title: A Phase II Trial of Hypofractionated Radiation Therapy for Prostate Cancer With High Risk Features After Radical Prostatectomy
Brief Title: Hypofractionated Radiation Therapy for Treating Prostate Cancer High-Risk Features Following Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1754; NCI-2018-00943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1754 (Other: Mayo Clinic); 17-009199 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-06-05; First posted 2018-06-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Prostate Adenocarcinoma; Stage IIB Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (hypofractionated radiation therapy) (Experimental): Participants undergo hypofractionated radiation therapy over 15-30 minutes every other day over 2 weeks, for 5 treatments.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (radiation therapy, androgen suppression therapy) (Experimental): Beginning 8-10 weeks before radiation therapy, participants receive androgen suppression therapy SC or IM for up to 6 months (at the discretion of the treating physician). Participants then undergo hypofractionated radiation therapy as Group I.
  Interventions: Drug: Androgen Suppression; Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (radiation therapy, androgen suppression therapy) (Experimental): Participants receive androgen suppression therapy as Group II for up to 18 months (at the discretion of the treating physician), then undergo hypofractionated radiation therapy over 15-30 minutes every other day over 1-2 weeks, for 1-5 treatments.
  Interventions: Drug: Androgen Suppression; Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Androgen Suppression — Given androgen suppression therapy
  Other Names: Androgen Ablation; androgen deprivation
  Arms: Group II (radiation therapy, androgen suppression therapy); Group III (radiation therapy, androgen suppression therapy)
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well hypofractionated radiation therapy works in treating participants with prostate cancer high-risk features following radical prostatectomy. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if stereotactic body radiation therapy (SBRT) would result in similar freedom from failure (FFF) than standard fractionation photon therapy.

EXPLORATORY OBJECTIVES:

I. After completion of radiation therapy, determine the incidence of grade 2 or greater genitourinary (GU) and gastrointestinal (GI) toxicity at 6 months (Common Terminology Criteria for Adverse Events [CTCAE] version 4).

II. After completion of radiation therapy, determine the incidence of grade 3 or greater GU and GI toxicity at 6 months (CTCAE version 4).

III. After completion of radiation therapy, determine the incidence of quality of life issues following completion of radiation therapy.

IV. After completion of radiation therapy, determine the incidence of impotence after the use of radiation therapy at 3 years.

V. After completion of radiation therapy, determine the incidence of freedom from biochemical failure (FFBF) at 5 years.

VI. After completion of radiation therapy, determine the incidence of clinical failure: local and/or distant at 5 years.

VII. After completion of radiation therapy, determine the incidence of salvage androgen deprivation use (SAD) at 5 years.

VIII. After completion of radiation therapy, determine the incidence of progression free survival: using clinical, biochemical and SAD as events at 5 years.

IX. After completion of radiation therapy, determine the incidence of overall survival at 5 years.

X. After completion of radiation therapy, determine the incidence of disease-specific survival at 5 years.

XI. Determine the impact of radiation therapy on quality of life. XII. Determine overall GI and GU toxicity. XIII. Determine prostate and normal structure movement during radiation therapy (RT) with the use of scans.

XIV. Correlate pathologic and radiologic findings with outcomes. XV. Correlate pre-RT prostate specific antigen (PSA) levels with outcomes. XVI. Correlate variation in proton therapy or x-ray dosimetry and outcomes. XVII. Develop a quality assurance process for prostate proton therapy. XVIII. Prospectively collect information that will help to define dose-volume relationships of normal structures with acute and chronic toxicity.

XIX. Allow for future research of pathologic risk factors that may influence prognosis; this information will help us to attempt to characterize their presence in prostate cancer with high risk features after prostatectomy and their potential effect on outcomes.

XX. Possibly compare dosimetric parameters of an IMRT plan with the proton therapy radiation plan.

OUTLINE: Participants are assigned to 1 of 3 groups.

GROUP I: Participants undergo hypofractionated radiation therapy over 15-30 minutes every other day over 2 weeks, for 5 treatments.

GROUP II: Beginning 8-10 weeks before radiation therapy, participants receive androgen suppression therapy subcutaneously (SC) or intramuscularly (IM) for up to 6 months (at the discretion of the treating physician). Participants then undergo hypofractionated radiation therapy as Group I.

GROUP III: Participants receive androgen suppression therapy as Group II for up to 18 months (at the discretion of the treating physician), then undergo hypofractionated radiation therapy over 15-30 minutes every other day over 1-2 weeks, for 1-5 treatments.

After completion of study treatment, participants are followed up at 3 and 12 months, annually for 4 years, then every 2 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma at the time of surgery
* Pathologic stages T2-T3b, N0-Nx-N1, M0-1 as staged by the pathology report (American Joint Committee on Cancer [AJCC] criteria 8th edition [Ed.])
* One or more high risk features including: seminal vesicle invasion, extracapsular extension, positive margins, or a PSA post surgery between 0.2 and < 2.0
* PSA values < 2 ng/ml within 90 days prior to enrollment. Obtained at least 6 weeks after surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 assessed within 90 days of enrollment
* Patients must sign Institutional Review Board (IRB) approved study specific informed consent
* Patients must complete all required pre-entry tests within the specified time frames
* Patients must be able to start treatment (androgen suppression [AS] or radiation) within 120 days of study registration
* Members of all races and ethnic groups are eligible for this trial
* Patients from outside of the United States may participate in the study

Exclusion Criteria:

* Previous pelvic radiation
* Prior androgen suppression therapy for prostate cancer for more than 6 months
* Active rectal diverticulitis, Crohn's disease affecting the rectum or ulcerative colitis (non-active diverticulitis and Crohn's disease not affecting the rectum are allowed)
* Prior systemic chemotherapy for prostate cancer
* History of proximal urethral stricture requiring dilatation
* Current and continuing anticoagulation with warfarin sodium (coumadin), heparin, low- molecular weight heparin, Clopidogrel bisulfate (plavix), or equivalent (unless it can be stopped to manage treatment related toxicity, to have a biopsy if needed, or place markers)
* Major medical, addictive or psychiatric illness which in the investigator's opinion, will prevent the consent process, completion of the treatment and/or interfere with follow-up. (Consent by legal authorized representative is not permitted for this study)
* Evidence of any other cancer within the past 5 years and < 50% probability of a 5 year survival. (Prior or concurrent diagnosis of basal cell or non-invasive squamous cell cancer of the skin is allowed)
* History of myocardial infarction or decompensated congestive heart failure (CHF) within the last 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Freedom from failure (FF) | Up to 5 years
  Will be defined as the first occurrence of clinical failure (local recurrence, regional recurrence, or distant metastasis), the start/re-start of salvage therapy including androgen suppression, and biochemical failure (PSA >= 0.5 ng/ml).

OTHER OUTCOMES:
Development of quality assurance process for prostate proton therapy | Up to 5 years
Overall survival at 5 years | Up to 5 years
  Overall survival is defined as the time from enrollment until death due to any cause.
Freedom from biochemical failure (FFBF) | Up to 5 years
  Biochemical failure is defined as a rise in prostate-specific antigen (PSA) levels after treatment, indicating that the cancer may be recurring or progressing.
Disease-free survival | Up to 5 years
  Will be estimated with a Kaplan-Meier estimator and curve. Estimates will be given for specific time points along with 95% CIs.
Progression free survival | Up to 5 years
  Will use clinical, biochemical and SAD as events. Will be estimated with a Kaplan-Meier estimator and curve. Estimates will be given for specific time points along with 95% CIs.
Salvage androgen suppression use at 5 years | Up to 5 years following completion of radiation therapy
  Will be assessed by the number of patients using salvage androgen deprivation use (SAD) at 5 years post radiation therapy
Impotence at 3 years | Up to 3 years after completion of radiation therapy
  Summation of relative scores for sexual function items (items 31 through 39) from the Expanded Prostate Cancer Index Composite (EPIC) instrument will be used to measure each individual's quality of life. The EPIC questionnaire is designed to measure Quality of Life issues in patients with Prostate Cancer. The questionnaire consists of 32 questions in 5 domains. Each question is answered on a 5-point scale such as 0-4 where 1=no problem and 4=big problem.
Quality of life (QOL) | Up to 5 years
  Summation of relative scores for quality of life items from the Expanded Prostate Cancer Index Composite (EPIC) instrument will be used to measure each individual's quality of life. The EPIC questionnaire is designed to measure Quality of Life issues in patients with Prostate Cancer. The questionnaire consists of 32 questions in 5 domains. Each question is answered on a 5-point scale such as 0-4 where 1=no problem and 4=big problem.
Distant metastasis | Up to 5 years
  Distant metastasis is cancer that has spread from the original (primary) tumor location to distant organs or distant lymph nodes.
Local/distant failure | Start of treatment assessed up to 5 years
  Will be measured from the treatment start date to the date of documented local failure as determined either by clinical exam, imaging, or by prostate re-biopsy.
Grade 2 or higher and grade 3 or higher GI and GU toxicity | 3 years
  Will be performed using NCI CTCAE v4 criteria. The maximum grade for each type of acute adverse events (AE) will be recorded for each patient.
Acute grade 2 or higher and grade 3 or higher genitourinary (GU) and gastrointestinal (GI) toxicity | Up to 5 years
  Assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 criteria. The maximum grade for each type of acute adverse events (AE) will be recorded for each patient.
Pathologic and radiologic findings | Up to 5 years
  Correlated with outcome.
Estimation of prostate and normal structure movement | Up to 5 years
Dose volume relationship of normal structures with toxicity | Up to 5 years
Potentially, future research of pathologic risk factors | Up to 5 years
Possible comparison of an intensity-modulated radiation therapy (IMRT) plan with the proton therapy radiation plan | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E. Vargas, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials